CLINICAL TRIAL: NCT00332956
Title: A Phase 2 (a), Dose-Blinded, Block-Randomized, Dose and Schedule Selection Study to Evaluate the Immunogenicity and Safety of the Recombinant Plague Vaccine rF1V in Healthy Volunteers
Brief Title: Title: Recombinant Plague Vaccine rF1V in Healthy Volunteers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: DynPort Vaccine Company LLC, A GDIT Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: rF1V-02(a)
Record Dates: First submitted 2006-06-01; First posted 2006-06-02 (Estimated); Last update posted 2011-12-02 (Estimated); Status verified 2011-11

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Group 1 (Active Comparator): Volunteers will be vaccinated with 80 mcg rF1V vaccine on Study Days 0 , 28, 182
  Interventions: Biological: rFIV vaccine
- Group 2 (Active Comparator): Volunteers will be vaccinated with 80 mcg of rF1V vaccine at Study Days 0, 56, 182
  Interventions: Biological: rF1V vaccine
- Group 3 (Active Comparator): Volunteers will be vaccinated with 160 mcg rF1V vaccine given on Study Days 0, 28, 182
  Interventions: Biological: rF1V vaccine
- Group 4 (Active Comparator): Volunteers will be vaccinated with 160 mcg rf1V vaccine on Study Days 0, 56, 182
  Interventions: Biological: rF1V vaccine 160 mcg given on Study Days 0, 56, 182

INTERVENTIONS:
Biological: rFIV vaccine — rF1V vaccine 80 mcg given by intramuscular (IM) injection into the arm on study Days 0, 28, 182
  Other Names: Recombinant Plague Vaccine rF1V
  Arms: Group 1
Biological: rF1V vaccine — rF1V 80 mcg vaccine given by intramuscular (IM) injection into the arm on study Days 0, 56, 182
  Other Names: Recombinant Plague Vaccine rF1V
  Arms: Group 2
Biological: rF1V vaccine — rF1V 160 mcg vaccine given by intramuscular (IM) injection into the arm on Study Days 0, 28, 182
  Other Names: Recombinant Plague Vaccine rF1V
  Arms: Group 3
Biological: rF1V vaccine 160 mcg given on Study Days 0, 56, 182 — rF1V 160 mcg vaccine given by Intramuscular (IM) injection into the arm on Study days 0. 56, 182
  Other Names: Recombinant Plague Vaccine rF1V
  Arms: Group 4

SUMMARY:
This Phase 2(a) clinical trial is designed as a dose-blinded, block-randomized, multi-center study to select a dosage and schedule of rF1V vaccine for further studies based on the immune response up to Day 210. Additional immunogenicity and safety/reactogenicity data will be collected through Day 540. Selection of dosage and schedule will be based on GMCs and seroconversion rates for anti-F1, anti-V and anti-rF1V antibody titers. Approximately 400 healthy adult volunteers will be enrolled (100 per group) in this study.

DETAILED DESCRIPTION:
Primary Objective: To select a dosage and schedule of rF1V vaccine for further study based on the immune response to F1 and V antigens up to Day 210.

Secondary Objectives: 1) To assess the safety of three injections of rF1V vaccine administered IM at two dosage levels.

2) To assess the onset and duration of the humoral immune response to F1 and V antigens.

3) To assess the humoral immune response to rF1V antigen. 4) To collect and store blood samples for future plague related research.

Exploratory Objectives:

To assess additional humoral immune responses to rF1V vaccine antigens.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female age 18 to 55 years
2. In good health
3. Acceptable ranges for the laboratory parameters
4. Normal ECG. If a volunteer is reported to have a benign ECG abnormality(e.g., sinus bradycardia) the results may be discussed with the medical monitors for the study.
5. Willing to have his/her blood samples stored for future plague research studies.
6. Signed the ICF and HIPPA and successfully completed the Test of Understanding (90% correct).
7. Agrees not to donate blood until at least 90 days following the last vaccination.
8. Volunteer is willing to comply with the requirements of the protocol through the post-vaccination Day 540 visit.
9. Female volunteers must be of non-childbearing potential or must not be pregnant. Must use 2 types of acceptable for of FDA approved contraception or abstinent.

Exclusion Criteria:

1. A history of plague disease or have previously received any plague vaccine.
2. Active tuberculosis or other systemic infectious process.
3. History of allergy to kanamycin or other aminoglycosides (e.g., gentamicin, tobramycin, amikacin)
4. Positive prescreening for human immunodeficiency virus (HIV); hepatitis C virus (HCV) or hepatitis B surface antigen (HbsAg).
5. A history of immunodeficiency or chronic illness requiring continuous or frequent medical intervention, acute/chronic untreated conditions, autoimmune disease or use of immunosuppressive medications.
6. Chronic, severe or recurrent joint pain (4 or more occurrences per year) or arthritis of any type.
7. A positive result on a urine drug screen that tests for common substances of abuse such as amphetamines, barbiturates, benzodiazepines, cocaine, opiates and cannabinoids.
8. A previous diagnosis of any serious psychiatric disorder. For this purpose, serious psychiatric disorder is defined as illness requiring hospitalization within the previous 12 months; routine administration of more than one medication to control anxiety, mood or sleep disorder; or history of suicide attempt.
9. Receipt of any blood product or immune globulin in the previous 6 months.
10. Receipt of any investigational vaccine in the previous 6 months
11. Donation of blood within 56 days prior to first vaccination or at any time prior to Day 210 visit.
12. Receipt of any investigational drug therapy within 30 days before the first dose of rF1V or intent to receive any other investigational drug therapy before the post-vaccination Day 540 visit.
13. A clinically significant abnormality on the ECG.
14. A body mass index > or equal to 35 kg/m2
15. Acute illness, evidence of significant active infection or systemic disease at time of enrollment that in the opinion of the Investigator would place the volunteer at an unacceptable risk for injury.
16. Personal history of multiple sclerosis, since immune system stimulation may exacerbate this disorder.
17. Occupational or other responsibilities that would prevent completion of participation in the study.
18. Licensed vaccines are not exclusionary but should be given at least 2 weeks before or after immunization (if live vaccine, 60 days before or after immunization) to avoid potential confusion of adverse reactions.
19. Screening laboratory values not within acceptable ranges.
20. A history of anaphylaxis or other serious adverse reactions to vaccines.
21. The female volunteer is pregnant
22. Receipt of therapy with immunosuppressive agents, including high-dose systemic corticosteroids (i.e., prednisone-equivalent dose of > or equal to 20 mg/day), within 3 months prior to or during the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 400 (Actual)
Dates: Start 2006-05; Primary Completion 2008-02 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
To select a final dosage and schedule of rF1V vaccine based on the immune response to F1 and V antigens up to Day 210 | Day 210 Interim Analysis

SECONDARY OUTCOMES:
To access the safety of three injections of rF1V vaccine administered IM at two dosage levels. | Day 210 Interim Analysis
To access the onset and duration of the humoral immune response to F1 and V antigens | Final Clinical Study Reort
To assess the humoral immune response to rF1V antigen | Final Clinical Study Report
To collect and store blood samples for future plague related research. | Through Study Day 540

CONTACTS AND LOCATIONS:
Overall Officials: Ivor Emmanual, MD, Principal Investigator — Benchmark Research; Steven Folkerth, MD, Principal Investigator — Clinical Research Center of Neveda; Richard Greenberg, MD, Principal Investigator — University of Kentucky - Department of Infectious Disease; Vicki Grieff, MD, Principal Investigator — Alta Clinical Research, LLC; John Jacobsen, MD, Principal Investigator — Meridian Clinical Research, LLC; Keith Reisinger, MD, Principal Investigator — Primary Physicians Research, Inc.; George Risi, MD, Principal Investigator — Infectious Disease Specialists, PC; L. Tyler Wadsworth, MD, Principal Investigator — Sundance Clinical Research; Iaasc Marcadis, MD, Principal Investigator — Palm Beach Research
Locations (9):
- United States (9):
  - Alta Clinical Research, LLC, Tucson, Arizona
  - Benchmark Research, San Francisco, California
  - Palm Beach Research, West Palm Beach, Florida
  - University of Kentucky - Dept. of Infectious Disease, Lexington, Kentucky
  - Sundance Clinical Research, St Louis, Missouri
  - Infectious Disease Specialists, PC, Missoula, Montana
  - Meridian clinical Research, LLC, Omaha, Nebraska
  - Clinical Research Center of Nevada, Las Vegas, Nevada
  - Primary Physicians Research, Inc., Pittsburgh, Pennsylvania